CLINICAL TRIAL: NCT07246811
Title: Rehabilitation Exercise Intervention for Rheumatoid Arthritis Patients Using Artificial Intelligence-Based Exercise Prescription System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-q003
Record Dates: First submitted 2025-08-11; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine Care Group (Active Comparator): Receives standardized RA disease management education and basic joint mobility exercises provided by rheumatology nurses.
  Interventions: Other: education and basic joint mobility exercises
- Paper Exercise Prescription Group (Active Comparator): Receives paper-based exercise prescription developed by rehabilitation therapists, including warm-up, formal training (bridging, modified bird-dog exercise, etc.) and cool-down stretching.
  Interventions: Other: paper-based exercise prescription
- AI Exercise Prescription Group (Experimental): Uses "Yidong Health AI Exercise Prescription System" delivered via WeChat mini-program, providing personalized exercise prescriptions (three sets: A/B/C) with AI Q&A module. Physicians adjust prescriptions weekly based on patient feedback.
  Interventions: Other: AI Exercise Prescription

INTERVENTIONS:
Other: AI Exercise Prescription — Uses "Yidong Health AI Exercise Prescription System" delivered via WeChat mini-program, providing personalized exercise prescriptions (three sets: A/B/C) with AI Q&A module. Physicians adjust prescriptions weekly based on patient feedback.
  Arms: AI Exercise Prescription Group
Other: education and basic joint mobility exercises — Receives standardized RA disease management education and basic joint mobility exercises provided by rheumatology nurses.
  Arms: Routine Care Group
Other: paper-based exercise prescription — Receives paper-based exercise prescription developed by rehabilitation therapists, including warm-up, formal training (bridging, modified bird-dog exercise, etc.) and cool-down stretching.
  Arms: Paper Exercise Prescription Group

SUMMARY:
This is a single-center, randomized, parallel-controlled trial evaluating the efficacy and safety of an artificial intelligence-based exercise prescription system for rehabilitation in rheumatoid arthritis (RA) patients. A total of 147 patients with low-to-moderate disease activity will be randomly assigned to three groups: AI exercise prescription group (personalized AI system guidance), paper exercise prescription group (traditional paper guidance), and routine care group. The intervention will last for 6 weeks with 6-month follow-up assessments evaluating joint function, pain, and quality of life indicators.

DETAILED DESCRIPTION:
This three-arm randomized controlled trial (RCT) uses Redcap system for 1:1:1 randomization. The AI exercise prescription group receives intervention through the "Yidong Health AI Exercise Prescription System" delivered via WeChat mini-program; the paper exercise prescription group receives traditional paper-based guidance; and the routine care group receives standardized health education and basic exercise instructions. The primary outcome measure is knee flexion range of motion (ROM) at 6 months, with secondary outcomes including HSS score, WOMAC index, TUG test, BBS balance scale, and other functional assessment measures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years Meets 2010 ACR/EULAR classification criteria for RA Low-to-moderate disease activity (assessed by rheumatologist) Knee joint involvement Willing and able to provide informed consent

Exclusion Criteria:

* Existing joint ankylosis (fibrous or bony) Acute flare or extra-articular soft tissue lesions Comorbid with other rheumatic diseases (e.g., SLE, Sjögren's syndrome) Severe hepatic or renal impairment Knee joint VAS pain score >4 (0-10 scale) Psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Knee flexion range of motion | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
  Knee Flexion Range of Motion Unit of Measure: Degrees (°) Knee flexion range of motion refers to the maximum angle through which the knee joint can bend, measured from the straight (extended) position to the farthest point the lower leg can move toward the thigh. This assessment evaluates the flexibility and functional mobility of the knee, which is critical for daily activities such as walking, climbing stairs, and sitting.
  Relevant definitions and criteria:
  A "normal" range of motion for knee flexion in adults is generally considered to be 135° to 150°, though this can vary slightly based on age, physical conditioning, and individual anatomy.
  Limited knee flexion (e.g., less than 90°) may indicate joint stiffness, muscle tightness, or underlying issues such as injury, arthritis, or post-surgical scarring.

SECONDARY OUTCOMES:
Hospital for Special Surgery (HSS) Score | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
  Hospital for Special Surgery (HSS) Score Unit of Measure: Points (out of 100) The Hospital for Special Surgery (HSS) Score is a comprehensive assessment tool used primarily in orthopedics, especially in evaluating the condition of the knee joint. It helps medical professionals determine the overall function and well - being of the knee, which is crucial for guiding treatment decisions, such as whether conservative management or surgical intervention is more appropriate.Total Score Range: The HSS Score ranges from 0 to 100 points.
  Interpretation of Scores:
  > 85 points: Considered "excellent". At this level, the knee is functioning very well, with minimal pain and good functional ability. In many cases, patients with such scores may not require significant medical intervention or may only need conservative measures like rest and exercise adjustments.
  70 - 85 points: Rated as "good". The knee has some minor issues, but overall function is still acceptable. Appropriate conservative
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
Timed Up and Go (TUG) Test | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
Berg Balance Scale (BBS) | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
Isokinetic Muscle Strength Test | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
Gait and Plantar Pressure Analysis | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
Arthritis Self-Efficacy Scale (ASES-8) | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
Patient Health Questionnaire-9 (PHQ-9) | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
Pittsburgh Sleep Quality Index (PSQI) | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
Health Assessment Questionnaire (HAQ) | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up
Laboratory indicators (RF, CRP, complete blood count) | Baseline, post-intervention (6 weeks), 3-month follow-up, 6-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT07246811/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT07246811/ICF_001.pdf